CLINICAL TRIAL: NCT03770481
Title: Using a Nurse-Led Communication Strategy to Improve Surrogates' Perception of Communication in the Intensive Care Unit
Brief Title: Using a Nurse-Led Communication Strategy for Surrogates in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Chiahui Chen, Principal Investigator, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 00008241
Record Dates: First submitted 2018-12-05; First posted 2018-12-10 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Communication Research
Keywords: communication; end-of-life; intensive care unit
MeSH Terms: conditions — Communication; Death

STUDY DESIGN:
Intervention Model Description: Two-groups comparison study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Assess the NLCS' feasibility (Experimental): Hypothesis: No significant differences will be observed in recruitment and attrition between NLCS intervention and control groups.
  Approach: Determine rates of enrollment and drop-outs between groups.
  Interventions: Behavioral: nurse-led communication strategy
- Assess the NLCS' acceptability (Experimental): Hypothesis: More surrogates agree that the NLCS is suitable, appropriate, effective and willing to adhere versus treatment as usual (TAU) communication.
  Approach: Assess outcome using the validated instrument, Client Satisfaction Questionnaire (CSQ-8).
  Interventions: Behavioral: nurse-led communication strategy
- Assess the NLCS' preliminary effects (Experimental): Hypothesis: NLCS improves communication and decreases surrogates' psychological distress (e.g., anxiety and depression) Approach: Compare pre- and post-intervention scores of the Quality of Communication (QOC) questionnaire, Hospital Anxiety and Depression Scale (HADS), and Decisional Conflict Scale (DCS) between intervention and control groups.
  Interventions: Behavioral: nurse-led communication strategy

INTERVENTIONS:
Behavioral: nurse-led communication strategy — Nurse-led communication strategy (NLCS) applies 'COMFORT' framework that research nurses use the framework to engage one communication session per day with surrogates and two discussions with bedside nurses or attending physician during the ICU stay.

SUMMARY:
Communication is one of the greatest health needs for high quality end-of-life (EOL) care in the intensive care unit (ICU), especially when patients are too ill to speak for themselves and rely on surrogates to make EOL decisions. Yet, there is no effective nursing intervention designed to improve communication between surrogates and clinicians. In order to enhance understanding of the surrogates' needs in the transition to EOL, this study will propose a new theory-grounded communication intervention, Nurse-Led Communication Strategy (NLCS) and will evaluate its feasibility, acceptability, and preliminary effects.

DETAILED DESCRIPTION:
Background: In 2014, 14.7% of Americans died using intensive care unit (ICU) services. It is a clinical imperative to provide high quality EOL care. Strong communication with surrogates is vital for high quality EOL care due to the fact that seriously ill patients often cannot talk, and they rely on surrogates (often family members) to make EOL decisions. There have been many studies conducted in the past, trying to improve EOL communication. Yet, evidence shows that communication remains poor in the ICU. To date, there is lack of evidence for a particular nursing strategy that effectively improves communication and the quality of EOL care in the ICU. The goal of this proposed study is to develop a new nurse-led communication strategy (NLCS). Specific Aim: To assess the NLCS's feasibility, acceptability, and preliminary effects among surrogates of patients who are unable to communicate in the ICU. Theory: NLCS is grounded in the state-of-the art framework "COMFORT" which has guided a validated and effective communication training for nurses in the care of patients with life-threatening illness and their families. NLCS applies 'COMFORT' into a usable nursing communication strategy that research nurses use the framework to engage one communication session per day with surrogates during the ICU stay. Methods: A single-center pilot two-groups comparison study. The study design involves the recruitment of surrogates in the ICU to evaluate the feasibility, acceptability, and preliminary effects of the NLCS. Analysis: To assess feasibility, we will use descriptive statistics and a COSORT (Consolidated Standards of Reporting Trials) flow diagram to determine recruitment and attrition. For acceptability, we will use an unpaired (independent) t test to compare the scores of the Client Satisfaction Questionnaire (CSQ-8)and between intervention and control groups. To evaluate preliminary effects of the intervention, we will compare the pre- and post-test scores of the Quality of Communication (QOC) questionnaire, Hospital Anxiety and Depression Scale (HADS), and Decisional Conflict Scale (DCS) between intervention and control groups. It determines whether the NLCS is perceived as appropriate, acceptable, and potentially effective. The by-product analysis uses a linear regression to determine which factors are associated with the scores of the . This proposal provides an opportunity for the first time to develop a theory-grounded nursing communication strategy that is feasible, acceptable, and poses low cognitive load for surrogates in the ICU, and it enhances the understanding of surrogates' needs in the transition to EOL and thereby potentially improves the quality of EOL care. This research training will take place at the University at Buffalo School of Nursing, an exceptional research-intensive university, under the mentorship of Dr. Chang and Dr. Lorenz (methodology), Dr. Sullivan (EOL studies), and Dr. Wittenberg (communication theory). The training plan will provide the investigator with research skills and the preliminary data.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  1. Age ≥ 18 years
  2. in the ICU for > 24 hours
  3. Mechanically ventilated within 24 hours of ICU admission
  4. Having an Acute Physiology and Chronic Health Evaluation (APACHE) IV ICU mortality prediction ≥ 20%
* Surrogates

  1. Age ≥ 18 years
  2. A legal New York State healthcare proxy documentation or A Family Health Care Decision Act (FHCDA) consent

Exclusion Criteria:

* Patients

  1. Decease or discharge from ICU within 24 hours
  2. Mechanically ventilated after 24 hours of ICU stay
  3. Able to communicate and make own decision
  4. Lack of a legal surrogate/proxy decision-maker to consent for patient participation
* Surrogates

  1. Lack of legal surrogate documentation
  2. Not able to complete consent process and questionnaires in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Rates of enrollment and drop-outs between intervention group (surrogates receive nurse-led communication strategy) and control group (surrogates receive treatment as usual communication) | During ICU stay, approximately 5 days
  Feasibility is measured by the number and timing of actual versus planned recruitment. Checklist is used to calculate the weekly recruitment rate which is the ratio of the enrollment out of the total number screened. The dropout rate is used to examine attrition of the intervention.
Scores of the Client Satisfaction Questionnaire (CSQ-8) between intervention group (surrogates receive nurse-led communication strategy) and control group (surrogates receive treatment as usual communication) | During ICU stay, approximately 5 days
  All participants will complete the Client Satisfaction Questionnaire (CSQ-8) at the time of ICU discharge to assess the acceptability of Nurse-Led Communication Strategy (NLCS) and Treatment as Usual (TAU) communication. The CSQ-8 include eight items assessing whether the intervention is perceived as appropriate, acceptable, and effective in improving communication in the ICU and whether participants are willing to participate if a similar study is offered. Their responses are scored from 1 to 4, and thus the possible total scores range from 8 to 32. Higher scores indicate greater satisfaction.
Pre- and post-intervention scores of the Quality of Communication (QOC) questionnaire between intervention group and control group. | During ICU stay, approximately 5 days
  The QOC has 13 items with two subscales (general communication skill and end-of-life scales). Each item score ranged from 0 to 10. Higher score of QOC indicated a more favorable perception of physician-family communication.
Pre- and post-intervention scores of the Hospital Anxiety and Depression Scale (HADS) between intervention group and control group. | During ICU stay, approximately 5 days
  The HADS is a 14-item/4-point Likert self-administered scale and consists of two subscales (depression and anxiety). The subscale total scores range from 0 (no distress) to 21 (severe distress), and a score above 11 indicates clinically significant symptoms of anxiety or depression.
Pre- and post-intervention scores of the Decisional Conflict Scale (DCS) between intervention group and control group. | During ICU stay, approximately 5 days
  The Decisional Conflict Scale has 10 items with three subscales: (a) uncertainty in choosing options, (b) factors influencing uncertainty in decision making, and (c) effective decision making. The Decisional Conflict Scale been frequently used among surrogate decision makers to evaluated decisional conflict or uncertainty. The score ranges from 0 (no decisional conflict) to 100 (extremely high decisional conflict).

CONTACTS AND LOCATIONS:
Locations (1):
- Buffalo General Medical Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350